CLINICAL TRIAL: NCT06517303
Title: Evaluation of the Implementation of Drug Prescription Recommendations Using Clinical Decision Support in Patients With Severe Obesity: Retrospective Study
Acronym: RECOB-MED
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200049; PREPS-19-127 (Other Grant/Funding Number: French ministry of health)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Obesity, Morbid; Drug Use
Keywords: prescription drug guidelines; clinical decision support system; Rule-based Alert System
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- retrospective study: Retrospective study of two data warehouses and the Delphi method

SUMMARY:
No drug prescription guidelines for severe obesity (BMI>35 kg/m2) are available, leading to non-standardized and / or potentially inappropriate drug management.

After validation of guidelines by the Delphi method, the main objective is to assess the agreement between the drug prescriptions and the guidelines after implementation in two health data warehouses.

The investigators will perform a retrospective, multicentric study in 2 hospitals. The investigators will check the relevance of rules (alerts) derived from the recommendations identified using the Delphi method.

DETAILED DESCRIPTION:
No drug prescription guidelines for severe obesity (BMI>35 kg/m2) are available, leading to non-standardized and / or potentially inappropriate drug management.

After validation of guidelines by the Delphi method, the main objective is to assess the agreement between the drug prescriptions and the guidelines after implementation in two health data warehouses.

The investigators will perform a retrospective, multicentric study in 2 hospitals. The investigators will check the relevance of rules (alerts) derived from the recommendations identified using the Delphi method.

The sponsor anticipate around 800 patients in the HEGP data warehouse and around 250 patients in the Rennes University Hospital data warehouse.

The main outcome will be the number of prescriptions concerned by rules, by type of recommendation, in patients with severe obesity.

Secondary outcomes will be :

1. Number of validated recommendations and their level of evidence,
2. Rate of prescriptions concerned by a computerized rule with pharmaceutical advice on the drug concerned by the rule. Sub-group analysis of this rate by type of recommendation.

The study will be conducted in 2 steps:

* Stage 1 (secondary endpoint): it consists of the final drafting of recommendations and submission to experts/analysis of feedback. This stage is scheduled to last 12 months.
* Stage 2 (primary and secondary judgment criteria): it consists of implementing the recommendations and studying the relevance of the rules. This stage is scheduled to last 8 months.

Around a hundred patients corresponding to this criteria will be extracted from the HEGP data warehouse

ELIGIBILITY:
Inclusion Criteria:

All patients aged 18 to 65 at the time of prescription with a BMI>35 kg/m² present in the clinical data warehouse of the HEGP and CHU Rennes during the study period with at least one hospitalization of more than 24h.

Exclusion Criteria:

* Patients who refused to have their records processed electronically.
* Patients with a history of bariatric surgery (sleeve gastrectomy, gastric band, gastric bypass) prior to hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 to 65 at the time of prescription with a BMI>35 kg/m² present in the clinical data warehouse
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-06-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
number of prescriptions concerned by rules, by type of recommendation | 8 months
  number of prescriptions concerned by rules, by type of recommendation, in patients with severe obesity.

SECONDARY OUTCOMES:
Number of validated recommendations and their level of evidence | 12 months
  Number of validated recommendations and their level of evidence, validated by experts
Rate of prescriptions concerned by a computerized rule with pharmaceutical advice on the drug concerned by the rule. | 8 months
  Rate of prescriptions concerned by a computerized rule with pharmaceutical advice on the drug concerned by the rule. Sub-group analysis of this rate by type of recommendation.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte SABATIER, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - HEGP, Paris
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. Data dictionary would be transmitted.
Supporting Information: Study Protocol
Time Frame: two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).